CLINICAL TRIAL: NCT05123508
Title: Treatment of Surgical Scars Following Breast Lifts/Reductions
Brief Title: Treatment of Breast Lift/Reduction Scars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCARCIP001
Record Dates: First submitted 2021-06-22; First posted 2021-11-17 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Scars
Keywords: Breast reduction scars; Breast lift scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Treatment arm and control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Arm (Experimental): 2940nm laser and BBL treatment
  Interventions: Device: 2940nm and BBL treatment
- Control Arm (Experimental): One side of the treatment area will act as a control. No treatment on the control side.
  Interventions: Other: Non-treatment side (Control)

INTERVENTIONS:
Device: 2940nm and BBL treatment — 2940nm and BBL treatment
  Arms: Treatment Arm
Other: Non-treatment side (Control) — No treatment
  Arms: Control Arm

SUMMARY:
Laser and light treatment for surgical scars following breast lifts/reductions

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate effectiveness of laser and light therapy for the treatment of surgical scars following breast lifts/reductions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects between 25 to 60 years of age inclusive
2. Fitzpatrick skin type I-IV
3. Subjects with post-surgical breast lift/reduction scar
4. A maximum of 8-10 weeks since surgery
5. Healed surgery wound in the treatment area
6. Willing to have photographs taken of the treatment area
7. Can read, understand and sign informed consent form (English only)
8. Has indicated willingness to participate in the study by signing an informed consent form
9. Agrees to adhere to the treatment and follow-up schedule and post treatment care instructions

Exclusion Criteria:

1. Fitzpatrick skin type V-VI
2. Breast reconstruction with radiation treatment
3. Is pregnant and/or lactating
4. Has tattoos, dysplastic nevi in the treatment area
5. History or current photosensitivity
6. History or current use of medication with photosensitizing properties within past 6 months
7. History or current of chronic reoccurring skin disease or disorder affecting treatment area
8. History or current cancer of any type
9. Has hormonal disorder
10. Has signs of actinic bronzing
11. Has open lacerations, and abrasions on the treatment area
12. History of keloid formation, or hypertrophic scar formation, or poor wound healing
13. History of bleeding disorder, or is currently taking anticoagulation medications
14. Has significant concurrent illnesses (controlled or uncontrolled), such as diabetes, lupus, epilepsy, or cardiac disorders, which might be aggravated as a result of treatment
15. Has participated in any clinical trial involving an investigational drug, device or cosmetic product or procedure within the past 30 days
16. The investigator feels that for any reason the subject is not eligible to participate in the study.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Improvement in surgical scars | 3 months
  Degree of improvement in scars using photographs assessed via modified Vancouver scar scale

SECONDARY OUTCOMES:
Overall improvement | 3 months
  The Patient and Observer Scar Scale (POSAS)
Overall Improvement | 3 months
  Global Aesthetic Improvement Scale (GAIS)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Cohen, MD, Principal Investigator — AboutSkin Research, LLC; Jason Pozner, MD, Principal Investigator — Sanctuary Plastic Surgery
Locations (2):
- United States (2):
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Sanctuary Plastic Surgery, Boca Raton, Florida